CLINICAL TRIAL: NCT02965300
Title: The Value of VOCs Analysis in Exhaled Breath for Pulmonary Benign and Malignant Lesion Diagnosis
Acronym: VOCs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Liang_An, MD,PHD, Chinese PLA General Hospital
Other Study IDs: S2016-110-01
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Lung Neoplasm; Lung Disease
Keywords: Pulmonary lesion; Volatile Organic Compositions(VOCs)
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Primary lung cancer: patients newly diagnosed with lung cancer by tissue biopsy and did not receive any treatment aiming at the tumor, including chemotherapy and radiotherapy.
- Benign lung lesion: Patients diagnosed with pulmonary benign diseases.
- Healthy control: Patients without any pulmonary abnormal symptoms or diseases

SUMMARY:
The purpose of this study is to analysis the volatile organic gases(VOCs) in exhaled breath of pulmonary lesion patients and healthy controls, in order to find the difference of composition and concentration among groups.

DETAILED DESCRIPTION:
Collect the exhaled gas in pulmonary lesion patients and healthy controls, using proton transfer reaction mass spectrometry to analysis the different composition and concentration of VOCs, to find the biomarker gases of distinguishing benign and malignant lesion of lung among different groups， and try to build a diagnostic model for lung lesion.

ELIGIBILITY:
Inclusion Criteria:

* cohort 1 :

Inclusion criteria:

Patients newly diagnosed with primary lung cancer by tissue biopsy and did not receive any treatment aiming at the tumor, including chemotherapy and radiotherapy.

Age ≥ 18 years

* cohort 2： Inclusion criteria： Patients diagnosed with pulmonary benign lesion by tissue biopsy or other examination.

Age ≥ 18 years

Exclusion Criteria:

patients who have more than one type of carcinoma patients diagnosed type 2 diabetes mellitus patients diagnosed chronic renal failure patients diagnosed upper digestive tract ulcer patients who reject to sign the informed consent from

* cohort 3： Healthy controls Volunteers without diagnosed lung diseases and pulmonary symptoms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung disease or healthy controls without lung diseases， and can cooperate with the collection of exhaled breath.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Mass-to-charge Ratio | 6 months
  It is the measurement result of VOCs in exhaled breath using PTR-MS device.

CONTACTS AND LOCATIONS:
Overall Officials: liang-an Chen, MD,PHD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- department of respiratory department ,Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
considering of personal privacy, the research-related individual participant data do not intend for public sharing.